CLINICAL TRIAL: NCT06029192
Title: Diastolic Function in Myotonic Dystrophy Type 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Abdallah FAYSSOIL, Associate Professor, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: ECHO-DM1
Record Dates: First submitted 2023-07-21; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Diastolic Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myotonic dystrophy type 1 (DM1) is a neuromuscular disorder in relation with an unstable expansion of CTG repeat. Patients with DM1 are at risk of arrhythmia and conduction disorders. Mortality are mainly related to respiratory failure and sudden death. Patients with DM1 may suffer from obesity, arterial hypertension, diabetes mellitus and sleep apnea. These comorbidities are classically associated with left ventricular diastolic dysfunction (DD) .

The investigators aim to assess the prevalence of left ventricular diastolic dysfunction in patients with myotonic dystrophy type 1 , the distribution of DD grading as well as the long-term prognosis of DM1 patients with a left ventricular diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* patients with genetic proven myotonic dystrophy type 1
* who experienced a Doppler- Echocardiography including an assessment of the left ventricular diastolic function

Exclusion Criteria:

* wall motion basal abnormalities
* significant valvular disease

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with myotonic dystrophy type 1 followed in a tertiary reference center.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 7 years

SECONDARY OUTCOMES:
Incidence of arrhythmia | 7 years
acute heart failure | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah FAYSSOIL, MD PhD, Principal Investigator — CHU Raymond Poincare
Locations (1):
- Hopital Raymond Poincare, Garches, France

IPD SHARING:
Plan to Share IPD: No